CLINICAL TRIAL: NCT00000309
Title: Serotonin/Dopamine Antagonism of Cocaine Effect
Brief Title: Serotonin/Dopamine Antagonism of Cocaine Effect: 1 - 1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to recruit adequate number of subjects
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lawrence H. Price, Professor of Psychiatry and Human Behavior, Butler Hospital
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09330-1; R01DA009330 (NIH); R01-09330-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine abuse, cocaine addiction
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
The purpose of this study is to evaluate use of risperidone with cocaine abusers. Study measures incorporate an appropriate integration of behavioral and neurobiological indices.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1994-08; Primary Completion 2000-01 (Actual); Study Completion 2000-01 (Actual)

PRIMARY OUTCOMES:
Analog mood scales
POMS
EPS sx

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Price, M.D., Principal Investigator — Brown University
Locations (1):
- Brown University School of Medicine, Providence, Rhode Island, United States